CLINICAL TRIAL: NCT02646215
Title: Inspiratory Muscle Training in Ehlers Danlos Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EDS-IMT
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Ehlers Danlos

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiratory muscle training group (Active Comparator): Threshold inspiratory muscle training
  Interventions: Device: Threshold inspiratory muscle training
- Control group (No Intervention): No training

INTERVENTIONS:
Device: Threshold inspiratory muscle training — Inspiratory muscle training
  Arms: Inspiratory muscle training group

SUMMARY:
Evaluation of the effect of inspiratory muscle training in Ehlers Danlos patients

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis for Ehlers Danlos syndrome combining genetics and clinical examination
* no infectious exacerbation in the last four weeks

Exclusion Criteria:

* respiratory comorbidities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
inspiratory muscle strength measured by sniff nasal inspiratory pressure | 2 minutes

SECONDARY OUTCOMES:
walked distance measured by six minutes walking test | 6 minutes
lung function by spirometry | 5 minutes
anxiety by hospital anxiety depression scale | 2 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique universitaire Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No